CLINICAL TRIAL: NCT02465060
Title: Molecular Analysis for Therapy Choice (MATCH)
Brief Title: Targeted Therapy Directed by Genetic Testing in Treating Patients With Advanced Refractory Solid Tumors, Lymphomas, or Multiple Myeloma (The MATCH Screening Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NCI-2015-00054; NCI-2015-00054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131 (Other: ECOG-ACRIN Cancer Research Group); EAY131 (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Bladder Carcinoma; Breast Carcinoma; Cervical Carcinoma; Colon Carcinoma; Colorectal Carcinoma; Endometrial Carcinoma; Esophageal Carcinoma; Exocrine Pancreas Carcinoma; Gastric Carcinoma; Glioma; Head and Neck Carcinoma; Hematopoietic and Lymphoid Cell Neoplasm; Kidney Carcinoma; Liver Carcinoma; Lung Carcinoma; Lymphoma; Malignant Uterine Corpus Neoplasm; Malignant Uterine Neoplasm; Melanoma; Multiple Myeloma; Ovarian Carcinoma; Prostate Carcinoma; Rectal Carcinoma; Recurrent Bladder Carcinoma; Recurrent Breast Carcinoma; Recurrent Cervical Carcinoma; Recurrent Colon Carcinoma; Recurrent Colorectal Carcinoma; Recurrent Esophageal Carcinoma; Recurrent Gastric Carcinoma; Recurrent Glioma; Recurrent Head and Neck Carcinoma; Recurrent Liver Carcinoma; Recurrent Lung Carcinoma; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Malignant Uterine Corpus Neoplasm; Recurrent Melanoma; Recurrent Multiple Myeloma; Recurrent Ovarian Carcinoma; Recurrent Pancreatic Carcinoma; Recurrent Prostate Carcinoma; Recurrent Rectal Carcinoma; Recurrent Skin Carcinoma; Recurrent Thyroid Gland Carcinoma; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma; Skin Carcinoma; Thyroid Gland Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Glioma; Hematologic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Lung Neoplasms; Lymphoma; Uterine Neoplasms; Melanoma; Multiple Myeloma; Ovarian Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Thyroid Neoplasms | interventions — adavosertib; Afatinib; binimetinib; Biopsy; Specimen Handling; capivasertib; copanlisib; Crizotinib; dabrafenib; Dasatinib; defactinib; erdafitinib; AZD4547; ipatasertib; larotrectinib; Magnetic Resonance Spectroscopy; Nivolumab; osimertinib; palbociclib; pertuzumab; 2C4 antibody; GSK2636771; X-Rays; Nuclear Medicine Department, Hospital; relatlimab; Immunoglobulin G; Disulfides; sapanisertib; Sunitinib; 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; trametinib; omipalisib; Trastuzumab; CT-P6; PF-05280014; trastuzumab biosimilar HLX02; Ogivri; Ontruzant; Ado-Trastuzumab Emtansine; ulixertinib; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (38):
- Subprotocol A (EGFR activating mutation) (Experimental): Patients with EGFR activating mutation receive afatinib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients may also undergo ECHO or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.
  Interventions: Drug: Afatinib; Drug: Afatinib Dimaleate; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging
- Subprotocol B (HER2 activating mutation) (Experimental): Patients with HER2 activating mutation receive afatinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Afatinib; Drug: Afatinib Dimaleate; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol C1 (MET amplification) (Experimental): Patients with MET amplification receive crizotinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation and collection of blood samples throughout the study. Patients may undergo biopsy at screening, on study, and/or at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Crizotinib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Procedure: Radiologic Examination
- Subprotocol C2 (MET exon 14 deletion/mutation) (Experimental): Patients with MET exon 14 deletion or other mutations that disrupt exon 14 receive crizotinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy on study and undergo radiologic evaluation and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Crizotinib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Procedure: Radiologic Examination
- Subprotocol E (EGFR T790M or rare activating mutation) (Experimental): Patients with EGFR T790M or rare activating mutation receive osimertinib (AZD9291) PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, ECHO or multigated acquisition scan (MUGA) during screening, and biopsy and collection of blood samples on trial and at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Cytology Specimen Collection Procedure; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Multigated Acquisition Scan; Drug: Osimertinib; Procedure: Radiologic Examination
- Subprotocol F (ALK translocation) (Experimental): Patients with ALK translocation receive crizotinib PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol G (ROS1 translocation or inversion) (Experimental): Patients with ROS1 translocation or inversion receive crizotinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol H (BRAF V600E/R/K/D mutation) (Experimental): Patients with BRAF V600E/R/K/D mutation receive dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Drug: Dabrafenib; Drug: Dabrafenib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Subprotocol I (PIK3CA mutation) (Experimental): Patients with PIK3CA mutation without RAS mutation or PTEN loss receive taselisib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Taselisib
- Subprotocol J (HER2 amplification >= 7 copy numbers) (Experimental): Patients receive pertuzumab IV over 30-60 minutes and trastuzumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, ECHO at screening and end of treatment, and biopsy and collection of blood samples on trial and at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Procedure: Radiologic Examination; Biological: Trastuzumab
- Subprotocol K1 (FGFR amplification) (Experimental): Patients with FGFR amplification receive erdafitinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout study. Patients may also undergo blood sample collection and tumor biopsy throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Drug: Erdafitinib; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging
- Subprotocol K2 (FGFR mutation or fusion) (Experimental): Patients with FGFR mutation or fusion receive erdafitinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT or MRI, and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Drug: Erdafitinib; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging
- Subprotocol L (mTOR mutation) (Experimental): Patients with mTOR mutation receive sapanisertib PO daily on days 1-28. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Sapanisertib
- Subprotocol M (TSC1 or TSC2 mutation) (Experimental): Patients with TSC1 or TSC2 mutation receive sapanisertib PO daily on days 1-28. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Sapanisertib
- Subprotocol N (PTEN mutation or deletion and PTEN expression) (Experimental): Patients with PTEN mutation or deletion and PTEN expression receive PI3K-beta inhibitor GSK2636771 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: PI3K-beta Inhibitor GSK2636771
- Subprotocol P (PTEN loss) (Experimental): Patients with PTEN loss receive PI3K-beta inhibitor GSK2636771 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: PI3K-beta Inhibitor GSK2636771
- Subprotocol Q (HER2 amplification) (Experimental): Patients with HER2 amplification receive trastuzumab emtansine intravenously (IV) over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Biological: Trastuzumab; Biological: Trastuzumab Emtansine
- Subprotocol R (BRAF fusion or BRAF non-V600 mutation) (Experimental): Patients with BRAF fusion or BRAF non-V600 mutation receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Subprotocol S1 (NF1 mutation) (Experimental): Patients with NF1 mutation receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Subprotocol S2 (GNAQ or GNA11 mutation) (Experimental): Patients with GNAQ or GNA11 mutation receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Subprotocol T (SMO or PTCH1 mutation) (Experimental): Patients with SMO or PTCH1 mutation receive vismodegib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or nuclear study during screening, tumor biopsy on study and CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging; Drug: Vismodegib
- Subprotocol U (NF2 inactivating mutation) (Experimental): Patients with NF2 inactivating mutation receive defactinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Drug: Defactinib; Drug: Defactinib Hydrochloride; Other: Laboratory Biomarker Analysis
- Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation) (Experimental): Patients with cKIT exon 9, 11, 13, or 14 mutation receive sunitinib PO QD on days 1-28 of each cycle. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo ECHO or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging; Drug: Sunitinib Malate
- Subprotocol W (FGFR pathway aberrations) (Experimental): Patients with FGFR1-3 mutation or translocation receive FGFR Inhibitor AZD4547 PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Drug: Fexagratinib; Other: Laboratory Biomarker Analysis
- Subprotocol X (DDR2 S768R, I638F, or L239R mutation) (Experimental): Patients with DDR2 S768R, I638F, or L239R mutation receive dasatinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Drug: Dasatinib; Other: Laboratory Biomarker Analysis
- Subprotocol Y (Akt mutation) (Experimental): Patients with Akt mutation receive capivasertib PO BID on days 1-4, 8-11, 15-18, and 22-25. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capivasertib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol Z1A (NRAS mutation in codon 12, 13, or 61) (Experimental): Patients with NRAS mutation in codon 12, 13, or 61 receive binimetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol Z1B (CCND1, 2, or 3 amplification with Rb by IHC) (Experimental): Patients with CCND1, 2, or 3 amplification that have tumor Rb expression by IHC receive palbociclib PO QD for 21 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Palbociclib
- Subprotocol Z1C (CDK4 or CDK6 amplification and Rb protein) (Experimental): Patients with CDK4 or CDK6 amplification and tumor Rb protein receive palbociclib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Palbociclib
- Subprotocol Z1D (Loss of MLH1 or MSH2 by IHC) (Experimental): Patients with mismatch repair deficiency (loss of MLH1 or MSH2 by IHC) receive nivolumab IV over 30 minutes on days 1 and 15 for 4 cycles and then on day 1 every 28 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion) (Experimental): Patients with NTRK1, NTRK2, or NTRK3 gene fusion receive larotrectinib (LOXO-101) PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo biopsies and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Larotrectinib; Drug: Larotrectinib Sulfate; Procedure: Magnetic Resonance Imaging
- Subprotocol Z1F (PIK3CA mutation) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsies at screening and end of treatment as well as CT or MRI at baseline and repeated every 2 cycles for the first 26 cycles then every 3 cycles thereafter until progressive disease or start of another MATCH treatment step.
  Interventions: Procedure: Biopsy Procedure; Procedure: Computed Tomography; Drug: Copanlisib; Drug: Copanlisib Hydrochloride; Other: Cytology Specimen Collection Procedure; Procedure: Magnetic Resonance Imaging
- Subprotocol Z1G (PTEN loss) (Experimental): Patients with PTEN loss receive copanlisib IV over 1 hour on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Drug: Copanlisib Hydrochloride; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol Z1H (PTEN mutation) (Experimental): Patients with PTEN mutation receive copanlisib IV over 1 hour on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Drug: Copanlisib Hydrochloride; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol Z1I (BRCA1 or BRCA2 gene mutation) (Experimental): Patients with BRCA1 or BRCA2 gene mutation receive adavosertib PO QD for 5 days for 2 weeks. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Subprotocol Z1K (AKT mutation) (Experimental): Patients receive ipatasertib PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Drug: Ipatasertib; Other: Laboratory Biomarker Analysis
- Subprotocol Z1L (BRAF fusion, aberration or non-V600 mutation) (Experimental): Patients with a BRAF non-V600 mutation or BRAF fusion, or another BRAF aberration receive ulixertinib (BVD-523FB) PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Ulixertinib
- Subprotocol Z1M (LAG-3 expression >= 1%) (Experimental): Patients receive nivolumab IV over 30 minutes and relatlimab IV over 30 minutes on day 1.Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Biological: Relatlimab

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775
  Arms: Subprotocol Z1I (BRCA1 or BRCA2 gene mutation)
Drug: Afatinib — Given PO
  Other Names: BIBW 2992; BIBW-2992; BIBW2992
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol B (HER2 activating mutation)
Drug: Afatinib Dimaleate — Given PO
  Other Names: (2E)-N-(4-((3-Chloro-4-fluorophenyl)amino)-7-(((3S)-tetrahydrofuran-3-yl)oxy)quinazolin- 6-yl)-4-(dimethylamino)but-2-enamide bis(hydrogen (2Z)-but-2-enedioate); BIBW 2992MA2; BIBW2992 MA2; Gilotrif
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol B (HER2 activating mutation)
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi
  Arms: Subprotocol Z1A (NRAS mutation in codon 12, 13, or 61)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol C1 (MET amplification); Subprotocol C2 (MET exon 14 deletion/mutation); Subprotocol E (EGFR T790M or rare activating mutation); Subprotocol J (HER2 amplification >= 7 copy numbers); Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion); Subprotocol T (SMO or PTCH1 mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation); Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion); Subprotocol Z1F (PIK3CA mutation)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol C1 (MET amplification); Subprotocol C2 (MET exon 14 deletion/mutation); Subprotocol E (EGFR T790M or rare activating mutation); Subprotocol J (HER2 amplification >= 7 copy numbers); Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion); Subprotocol T (SMO or PTCH1 mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation); Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion)
Drug: Capivasertib — Given PO
  Other Names: AZD 5363; AZD-5363; AZD5363; Truqap
  Arms: Subprotocol Y (Akt mutation)
Procedure: Computed Tomography — Undergo computed tomography (CT)
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion); Subprotocol T (SMO or PTCH1 mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation); Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion); Subprotocol Z1F (PIK3CA mutation)
Drug: Copanlisib — Given IV
  Other Names: BAY 80 6946; BAY 80-6946; BAY 806946; BAY-80-6946; BAY806946; PI3K Inhibitor BAY 80-6946
  Arms: Subprotocol Z1F (PIK3CA mutation); Subprotocol Z1G (PTEN loss); Subprotocol Z1H (PTEN mutation)
Drug: Copanlisib Hydrochloride — Given IV
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
  Arms: Subprotocol Z1F (PIK3CA mutation); Subprotocol Z1G (PTEN loss); Subprotocol Z1H (PTEN mutation)
Drug: Crizotinib — Given PO
  Other Names: Alkixen; Crizocent; MET Tyrosine Kinase Inhibitor PF-02341066; PF 02341066; PF-02341066; PF-2341066; PF02341066; Xalkori
  Arms: Subprotocol C1 (MET amplification); Subprotocol C2 (MET exon 14 deletion/mutation); Subprotocol F (ALK translocation); Subprotocol G (ROS1 translocation or inversion)
Other: Cytology Specimen Collection Procedure — Optional correlative studies
  Other Names: Cytologic Sampling
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol B (HER2 activating mutation); Subprotocol C1 (MET amplification); Subprotocol C2 (MET exon 14 deletion/mutation); Subprotocol E (EGFR T790M or rare activating mutation); Subprotocol F (ALK translocation); Subprotocol G (ROS1 translocation or inversion); Subprotocol H (BRAF V600E/R/K/D mutation); Subprotocol I (PIK3CA mutation); Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion); Subprotocol L (mTOR mutation); Subprotocol M (TSC1 or TSC2 mutation); Subprotocol N (PTEN mutation or deletion and PTEN expression); Subprotocol P (PTEN loss); Subprotocol Q (HER2 amplification); Subprotocol R (BRAF fusion or BRAF non-V600 mutation); Subprotocol S1 (NF1 mutation); Subprotocol S2 (GNAQ or GNA11 mutation); Subprotocol T (SMO or PTCH1 mutation); Subprotocol U (NF2 inactivating mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation); Subprotocol W (FGFR pathway aberrations); Subprotocol X (DDR2 S768R, I638F, or L239R mutation); Subprotocol Y (Akt mutation); Subprotocol Z1A (NRAS mutation in codon 12, 13, or 61); Subprotocol Z1B (CCND1, 2, or 3 amplification with Rb by IHC); Subprotocol Z1C (CDK4 or CDK6 amplification and Rb protein); Subprotocol Z1D (Loss of MLH1 or MSH2 by IHC); Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion); Subprotocol Z1F (PIK3CA mutation); Subprotocol Z1G (PTEN loss); Subprotocol Z1H (PTEN mutation); Subprotocol Z1I (BRCA1 or BRCA2 gene mutation); Subprotocol Z1K (AKT mutation); Subprotocol Z1L (BRAF fusion, aberration or non-V600 mutation); Subprotocol Z1M (LAG-3 expression >= 1%)
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK 2118436; GSK 2118436A; GSK-2118436; GSK-2118436A; GSK2118436; GSK2118436A
  Arms: Subprotocol H (BRAF V600E/R/K/D mutation)
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
  Arms: Subprotocol H (BRAF V600E/R/K/D mutation)
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Subprotocol X (DDR2 S768R, I638F, or L239R mutation)
Drug: Defactinib — Given PO
  Other Names: PF-04554878; VS-6063
  Arms: Subprotocol U (NF2 inactivating mutation)
Drug: Defactinib Hydrochloride — Given PO
  Arms: Subprotocol U (NF2 inactivating mutation)
Procedure: Echocardiography Test — Undergo echocardiography (ECHO)
  Other Names: EC; Echocardiography
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol E (EGFR T790M or rare activating mutation); Subprotocol J (HER2 amplification >= 7 copy numbers); Subprotocol T (SMO or PTCH1 mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation)
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ 42756493; JNJ-42756493; JNJ42756493
  Arms: Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion)
Drug: Fexagratinib — Given PO
  Other Names: ABSK-091; ABSK091; AZD4547; FGFR Inhibitor AZD4547; KB-74810
  Arms: Subprotocol W (FGFR pathway aberrations)
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
  Arms: Subprotocol Z1K (AKT mutation)
Other: Laboratory Biomarker Analysis — Undergo molecular analysis
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol B (HER2 activating mutation); Subprotocol C1 (MET amplification); Subprotocol C2 (MET exon 14 deletion/mutation); Subprotocol E (EGFR T790M or rare activating mutation); Subprotocol F (ALK translocation); Subprotocol G (ROS1 translocation or inversion); Subprotocol H (BRAF V600E/R/K/D mutation); Subprotocol I (PIK3CA mutation); Subprotocol J (HER2 amplification >= 7 copy numbers); Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion); Subprotocol L (mTOR mutation); Subprotocol M (TSC1 or TSC2 mutation); Subprotocol N (PTEN mutation or deletion and PTEN expression); Subprotocol P (PTEN loss); Subprotocol Q (HER2 amplification); Subprotocol R (BRAF fusion or BRAF non-V600 mutation); Subprotocol S1 (NF1 mutation); Subprotocol S2 (GNAQ or GNA11 mutation); Subprotocol T (SMO or PTCH1 mutation); Subprotocol U (NF2 inactivating mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation); Subprotocol W (FGFR pathway aberrations); Subprotocol X (DDR2 S768R, I638F, or L239R mutation); Subprotocol Y (Akt mutation); Subprotocol Z1A (NRAS mutation in codon 12, 13, or 61); Subprotocol Z1B (CCND1, 2, or 3 amplification with Rb by IHC); Subprotocol Z1C (CDK4 or CDK6 amplification and Rb protein); Subprotocol Z1D (Loss of MLH1 or MSH2 by IHC); Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion); Subprotocol Z1G (PTEN loss); Subprotocol Z1H (PTEN mutation); Subprotocol Z1I (BRCA1 or BRCA2 gene mutation); Subprotocol Z1K (AKT mutation); Subprotocol Z1L (BRAF fusion, aberration or non-V600 mutation); Subprotocol Z1M (LAG-3 expression >= 1%)
Drug: Larotrectinib — Given PO
  Other Names: ARRY 470; LOXO 101; LOXO-101; LOXO101
  Arms: Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion)
Drug: Larotrectinib Sulfate — Given PO
  Other Names: ARRY 470 Sulfate; LOXO 101 Sulfate; LOXO-101 Sulfate; Vitrakvi
  Arms: Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion)
Procedure: Magnetic Resonance Imaging — Undergo magnetic resonance imaging (MRI)
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol K1 (FGFR amplification); Subprotocol K2 (FGFR mutation or fusion); Subprotocol T (SMO or PTCH1 mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation); Subprotocol Z1E (NTRK1, NTRK2 or NTRK3 gene fusion); Subprotocol Z1F (PIK3CA mutation)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Subprotocol E (EGFR T790M or rare activating mutation)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Subprotocol Z1D (Loss of MLH1 or MSH2 by IHC); Subprotocol Z1M (LAG-3 expression >= 1%)
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
  Arms: Subprotocol E (EGFR T790M or rare activating mutation)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991
  Arms: Subprotocol Z1B (CCND1, 2, or 3 amplification with Rb by IHC); Subprotocol Z1C (CDK4 or CDK6 amplification and Rb protein)
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; BCD-178; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar BCD-178; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; Pertuzumab Biosimilar TQB2440; Pertuzumab-dpzb; Poherdy; Rhumab 2C4; rhuMAb2C4; RO4368451; TQB 2440; TQB-2440; TQB2440
  Arms: Subprotocol J (HER2 amplification >= 7 copy numbers)
Drug: PI3K-beta Inhibitor GSK2636771 — Given PO
  Other Names: GSK-2636771; GSK2636771
  Arms: Subprotocol N (PTEN mutation or deletion and PTEN expression); Subprotocol P (PTEN loss)
Procedure: Radiologic Examination — Undergo radiologic evaluation
  Other Names: Radiologic Evaluation; Radiologic Exam
  Arms: Subprotocol C1 (MET amplification); Subprotocol C2 (MET exon 14 deletion/mutation); Subprotocol E (EGFR T790M or rare activating mutation); Subprotocol J (HER2 amplification >= 7 copy numbers)
Procedure: Radionuclide Imaging — Undergo nuclear study
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
  Arms: Subprotocol A (EGFR activating mutation); Subprotocol T (SMO or PTCH1 mutation); Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation)
Biological: Relatlimab — Given IV
  Other Names: BMS 986016; BMS-986016; BMS986016; Immunoglobulin G4, Anti-(human Lymphocyte Activation Gene-3 Protein) (Human Heavy Chain), Disulfide with Human Light Chain, Dimer
  Arms: Subprotocol Z1M (LAG-3 expression >= 1%)
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228
  Arms: Subprotocol L (mTOR mutation); Subprotocol M (TSC1 or TSC2 mutation)
Drug: Sunitinib Malate — Given PO
  Other Names: SU 011248; SU 11248; SU-011248; SU-11248; SU011248; SU11248; sunitinib; Sutent
  Arms: Subprotocol V (cKIT exon 9, 11, 13, or 14 mutation)
Drug: Taselisib — Given PO
  Other Names: GDC-0032; RO5537381
  Arms: Subprotocol I (PIK3CA mutation)
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212
  Arms: Subprotocol H (BRAF V600E/R/K/D mutation); Subprotocol R (BRAF fusion or BRAF non-V600 mutation); Subprotocol S1 (NF1 mutation); Subprotocol S2 (GNAQ or GNA11 mutation)
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; HLX 02; HLX-02; HLX02; Kanjinti; Ogivri; Ontruzant; PF 05280014; PF-05280014; PF05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac
  Arms: Subprotocol J (HER2 amplification >= 7 copy numbers); Subprotocol Q (HER2 amplification)
Biological: Trastuzumab Emtansine — Given IV
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO 132365; PRO-132365; PRO132365; RO5304020; T-DM1; TDM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate
  Arms: Subprotocol Q (HER2 amplification)
Drug: Ulixertinib — Give PO
  Other Names: BVD-523; VRT752271
  Arms: Subprotocol Z1L (BRAF fusion, aberration or non-V600 mutation)
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC 0449; GDC-0449; GDC0449; Hedgehog Antagonist GDC-0449
  Arms: Subprotocol T (SMO or PTCH1 mutation)

SUMMARY:
This phase II MATCH screening and multi-sub-trial studies how well treatment that is directed by genetic testing works in patients with solid tumors, lymphomas, or multiple myelomas that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and does not respond to treatment (refractory). Patients must have progressed following at least one line of standard treatment or for which no agreed upon treatment approach exists. Genetic tests look at the unique genetic material (genes) of patients' tumor cells. Patients with genetic abnormalities (such as mutations, amplifications, or translocations) may benefit more from treatment which targets their tumor's particular genetic abnormality. Identifying these genetic abnormalities first may help doctors plan better treatment for patients with solid tumors, lymphomas, or multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

STEP 0 (Screening): Patients undergo biopsy along with molecular characterization of the biopsy material for specific, pre-defined mutations, amplifications, or translocations of interest via tumor sequencing and immunohistochemistry. Consenting patients also undergo collection of blood samples for research purposes.

STEPS 1, 3, 5, 7 (Treatment): Patients are assigned to 1 of 38 treatment subprotocols based on molecularly-defined subgroup. (See Arms Section)

STEPS 2, 4, 6 (Screening): Patients experiencing disease progression on the prior Step treatment or who could not tolerate the assigned treatment undergo review of their previous biopsy results to determine if another treatment is available or undergo another biopsy. Patients may have a maximum of 2 screening biopsies and 2 treatments per biopsy.

STEP 8 (Optional Research): Consenting patients undergo end-of-treatment biopsy and collection of blood samples for research purposes.

Additionally, patients may undergo a computed tomography (CT) scan, magnetic resonance imaging, and/or radionuclide imaging throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR SCREENING BIOPSY (STEP 0)
* Patients must be >= 18 years of age. Because no dosing or adverse event data are currently available on the use of study investigational agents in patients < 18 years of age, children are excluded from this study
* Patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to registration; patients that are pregnant or breast feeding are excluded; a patient of childbearing potential is anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria:

  * Has achieved menarche at some point
  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse prior to study entry, for the duration of study participation, and for 4 months after completion of study; should a patient or partner of the patient become pregnant or suspect a pregnancy while participating in this study, the treating physician should be informed immediately
* Patients must have histologically documented solid tumors or histologically confirmed diagnosis of lymphoma or multiple myeloma requiring therapy and meet one of the following criteria:

  * Patients must have progressed following at least one line of standard systemic therapy and there must not be other approval/standard therapy available that has been shown to prolong overall survival (i.e. in a randomized trial against another standard treatment or by comparison to historical controls); patients who cannot receive other standard therapy that has been shown to prolong overall survival due to medical issues will be eligible, if other eligibility criteria are met; if the patient is currently receiving therapy, the clinician must have assessed that the current therapy is no longer benefitting the patient prior to enrolling on MATCH, regardless of whether it is considered standard OR
  * Patients for whose disease no standard treatment exists that has been shown to prolong overall survival
  * NOTE: No other prior malignancy is allowed except for the following:
  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* Patients must have measurable disease
* Patients must meet the criteria below

  * Tumor tissue for the confirmation of "rare variant" by the MATCH assay is to be submitted, preferably from the same time of collection as that used to determine patient candidacy for treatment arm assignment

    * Registration to Step 0 must occur after stopping prior systemic anti-cancer therapy. There is no specific duration for which patients must be off treatment prior to registration to Step 0, as long as all eligibility criteria are met
    * Patients may have received other non-targeted, immunotherapy or targeted treatment between the prior genetic testing at the outside lab and registration to Step 0. The decision to stop such treatment in favor of participation in MATCH, if no further clinical benefit is expected, is per the treating physician's discretion. Documentation of a lack of response to the prior treatment is not required in these cases
    * Patients with an applicable "rare variant" must be able to meet the eligibility criteria for the appropriate subprotocols within 4 weeks following notification of treatment assignment
    * Patient meets one of the following criteria:

      * Patient is a candidate for Z1M based on local Clinical Laboratory Improvement Act (CLIA) assessment of mismatch repair deficiency (MMRd) by immunohistochemistry (IHC) or microsatellite instability (MSI) status by polymerase chain reaction (PCR), adequate tumor tissue is available for submission for mandatory central screening IHC and the patient will be able to meet the eligibility criteria for Z1M within 4 weeks following notification of treatment assignment OR
      * The sites have received results from one of the designated outside laboratories indicating a "rare variant" that is an actionable Mutation of Interest (aMOI) for specific select subprotocols
  * NOTE: There is no particular window of time after receiving the sequencing report notification of potential eligibility from an outside lab in which the patient must be registered to Step 0, but treatment slots will be assigned on a first come, first serve basis to those who do register to Step 0, and are not held for those notified of potential eligibility who do not register to Step 0
  * NOTE: Treatment assignment (and the start of the associated deadline for Step 1 registration) may occur shortly after Step 0 registration. Note that certain "rare variant" arms require submission of archival tissue for central IHC testing to determine treatment assignment. For those arms, adequate tissue for the central IHC is required to be available for submission
  * NOTE: Other potential aMOIs that would be eligibility criteria for "NON RARE" arms, as determined by the designated laboratories, are not applicable for this process in MATCH
* Patient must not require the use of full dose coumarin-derivative anticoagulants such as warfarin; low molecular weight heparin is permitted for prophylactic or therapeutic use; factor X inhibitors are permitted

  * NOTE: Warfarin may not be started while enrolled in the EAY131 study
  * Stopping the anticoagulation for biopsy should be per site standard operating procedure (SOP)
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 1 and a life expectancy of at least 3 months
* Patients must not currently be receiving any other investigational agents
* Patients must not have any uncontrolled intercurrent illness including, but not limited to:

  * Symptomatic congestive heart failure (New York Heart Association [NYHA] classification of III/IV)
  * Unstable angina pectoris or coronary angioplasty, or stenting within 6 months prior to registration to Step 0, 2, 4, 6
  * Cardiac arrhythmia (ongoing cardiac dysrhythmias of National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]4 grade >= 2)
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Intra-cardiac defibrillators
  * Known cardiac metastases
  * Abnormal cardiac valve morphology (>= grade 2) documented by echocardiogram (ECHO) (as clinically indicated); (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study); subjects with moderate valvular thickening should not be entered on study
  * NOTE: To receive an agent, patient must not have any uncontrolled intercurrent illness such as ongoing or active infection; patients with infections unlikely to be resolved within 2 weeks following screening should not be considered for the trial
* Patients must be able to swallow tablets or capsules; a patient with any gastrointestinal disease that would impair ability to swallow, retain, or absorb drug is not eligible
* Patients who are human immunodeficiency virus (HIV)-positive are eligible if:

  * CD4+ cell count greater or equal to 250 cells/mm^3
  * If patient is on antiretroviral therapy, there must be minimal interactions or overlapping toxicity of the antiretroviral therapy with the experimental cancer treatment; for experimental cancer therapeutics with CYP3A/4 interactions, protease inhibitor therapy is disallowed; suggested regimens to replace protease inhibitor therapy include dolutegravir given with tenofovir/emtricitabine; raltegravir given with tenofovir and emtricitabine; once daily combinations that use pharmacologic boosters may not be used
  * No history of non-malignancy acquired immune deficiency syndrome (AIDS)-defining conditions other than historical low CD4+ cell counts
  * Probable long-term survival with HIV if cancer were not present
* Any prior therapy, radiotherapy (except palliative radiation therapy of 30 gray [Gy] or less), or major surgery must have been completed >= 4 weeks prior to start of treatment; all adverse events due to prior therapy have resolved to a grade 1 or better (except alopecia and lymphopenia) by start of treatment; palliative radiation therapy must have been completed at least 2 weeks prior to start of treatment; the radiotherapy must not be to a lesion that is included as measurable disease

  * NOTE: Prostate cancer patients may continue their luteinizing hormone-releasing hormone (LHRH) agonist
  * NOTE: For patients entering the study via the original screening process, patients may receive non-protocol treatment after biopsy (if clinically indicated) until they receive notification of results; however, lack of response must be documented prior to registration to Step 1; new non-protocol treatment will NOT be permitted as intervening therapy after registration to Step 0; the only intervening treatment permitted is prior therapy that the patient already received prior to Step 0 registration; the decision to stop the intervening non-protocol treatment will be left up to the treating physician if patient has an aMOI; however, patients will need to be off such therapy for at least 4 weeks before receiving any MATCH protocol treatment
  * NOTE: For patients entering the study via a designated outside laboratory, no intervening systemic non-protocol treatment is permitted after Step 0 registration; all other eligibility requirements still apply to these patients, including the washouts for prior therapy noted above in this section, the time restrictions outlined, and the eligibility criteria for the intended subprotocol
* Patients with brain metastases or primary brain tumors must have completed treatment, surgery or radiation therapy >= 4 weeks prior to start of treatment
* Patients must have discontinued steroids >= 1 week prior to registration to Step 0 and remain off steroids thereafter, except as permitted; patients with glioblastoma (GBM) must have been on stable dose of steroids, or be off steroids, for one week prior to registration to treatment (Step 1, 3, 5, 7)

  * NOTE: The following steroids are permitted (low dose steroid use is defined as prednisone 10 mg daily or less, or bioequivalent dose of other corticosteroid):

    * Temporary steroid use: e.g. for CT imaging in setting of contrast allergy
    * Low dose steroid use for appetite
    * Chronic inhaled steroid use
    * Steroid injections for joint disease
    * Stable dose of replacement steroid for adrenal insufficiency or low doses for non-malignant disease
    * Topical steroid
    * Steroids required to manage toxicity related to study treatment, as described in the subprotocols
    * Steroids required as pre- or post-chemotherapy medication for acceptable intervening chemotherapy

      * NOTE: Steroids must be completed alongside last dose of chemotherapy
* Leukocytes >= 3,000/mcL (within 2 weeks prior to screening step registration and within 4 weeks prior to treatment step registration)
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 2 weeks prior to screening step registration and within 4 weeks prior to treatment step registration)
* Platelets >= 100,000/mcL (within 2 weeks prior to screening step registration and within 4 weeks prior to treatment step registration)
* NOTE: Patients with documented bone marrow involvement by lymphoma are not required to meet the above hematologic parameters, but must have a platelet count of at least 75,000/mcL and neutrophil count of at least 1,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (unless documented Gilbert's syndrome, for which bilirubin =< 3 x institutional ULN is permitted) (within 2 weeks prior to screening step registration and within 4 weeks prior to treatment step registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (up to 5 times ULN in presence of liver metastases) (within 2 weeks prior to screening step registration and within 4 weeks prior to treatment step registration)
* Creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional ULN

  * As defined by the Cockcroft-Gault equation (within 2 weeks prior to screening step registration and within 4 weeks prior to treatment step registration)
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to registration to screening step and must meet the following cardiac criteria:

  * Resting corrected QT interval (QTc) =< 480 msec

    * NOTE: If the first recorded QTc exceeds 480 msec, two additional, consecutive ECGs are required and must result in a mean resting QTc =< 480 msec; it is recommended that there are 10-minute (+/- 5 minutes) breaks between the ECGs
  * The following only need to be assessed if the mean QTc > 480 msec

    * Check potassium and magnesium serum levels
    * Correct any identified hypokalemia and/or hypomagnesemia and may repeat ECG to confirm exclusion of patient due to QTc
    * For patients with heart rate (HR) 60-100 beats per minute (bpm), no manual read of QTc is required
    * For patients with baseline HR < 60 or > 100 bpm, manual read of QT by trained personnel is required, with Fridericia correction applied to determine QTc
    * Patient must not have hypokalemia (value < institutional lower limit of normal)
  * No factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval

    * NOTE: Patient must be taken off prohibited medication prior to registration to the screening step (Step 0, 2, 4, 6) and remain off these medications thereafter, unless permitted on a subprotocol for the management of treatment related toxicity; patient must be off the drug for at least 5 half-lives prior to registration to the treatment step (Step 1, 3, 5, 7); the medication half-life can be found in the package insert for Food and Drug Administration (FDA) approved drugs
* ELIGIBILITY CRITERIA FOR FIRST TREATMENT (STEP 1)
* NOTE: For patients entering step 0 with assay results from outside laboratories, no systemic treatment is allowed after step 0 registration
* As MATCH is designed to add additional subprotocols, implement limited expansions of accrual for certain subprotocols, and/or amend existing arm-specific eligibility criteria, some patients entering under the original screening method may be eligible to have their results rerun in MATCHbox, even if they did not match to a treatment initially or did not receive a treatment assignment due to a lack of available assignment slots; patients whose sequence results will be rerun through MATCHbox must also meet the following criteria:

  * Samples must have been collected within 5 months of the activation of the addendum, as there is an additional month needed to get the patients on trial
  * Patient has not had treatment within the 5 months that resulted in a PR or better after the performance of the screening assessment
  * Patient must meet eligibility criteria, including performance status 1 or better and life expectancy of at least 3 months
  * Patients must meet the eligibility requirements with the following exceptions:

    * Patients may have received other non-targeted, immunotherapy or targeted treatment, which could be stopped in favor of returning to MATCH, if no response to the interim treatment has occurred and no further benefit is expected from this interim treatment, per the treating physician's discretion; documentation of a lack of response to the interim treatment is not required in these cases; however, the following restrictions apply:

      * Enrollment onto another investigational therapeutic study is not permitted
      * Patient cannot be responding to interim treatment, since the benefit of the MATCH treatment is unknown and may deprive patient of an effective treatment if it were given when a patient is responding to another treatment
  * NOTE: Patients meeting these criteria will NOT be biopsied at this time point; instead, their step 0 results will be re-interrogated to determine if another treatment is available
* ELIGIBILITY CRITERIA FOR SECOND SCREENING (STEP 2)
* Patient's disease has progressed on Step 1 treatment or patient could not tolerate assigned treatment

  * NOTE: PATIENTS ENTERING STEP 1 WITH A "RARE VARIANT" FROM AN "OUTSIDE" LAB ARE NOT ELIGIBLE FOR STEP 2
* No response and progression (or inability to tolerate further treatment) occurred < 6 months from start of step 1 treatment

  * NOTE: Patients meeting these criteria will NOT be biopsied at this time point; instead, their step 0 MATCH assay results will be re-interrogated to determine if another treatment is available upon registration to this study step; it is not necessary to confirm the availability of another potential treatment assignment in advance; only aMOIs detected by the MATCH assay may be used for the determination of eligibility to a relevant subprotocol OR
* Progression (or inability to tolerate further treatment) occurred after a (1) response OR (2) after >= 6 months from start of step 1 treatment; patient must have tumor amenable to percutaneous biopsy and be willing and able to undergo a tumor biopsy or bone marrow aspirate for collection and submission of tumor tissue OR patient will be undergoing a procedure due to medical necessity during which the tissue may be collected for the central determination of the presence of one or more of the specific "actionable" mutations/amplifications of interest (aMOI); archived specimens cannot be accepted
* Patients must meet eligibility criteria as defined in step 0
* Patient must not have been assigned to step 1 treatment based on a "rare variant" determined by a designated outside laboratory
* ELIGIBILITY CRITERIA FOR SECOND TREATMENT (STEP 3)
* NOTE: If screening biopsy samples were submitted during step 2, patients may receive non-protocol treatment after biopsy (if clinically indicated) until they receive notification of results however, lack of response must be documented prior to registration to step 3; new non-protocol treatment will NOT be permitted as intervening therapy after registration to step 2; the decision to stop the intervening nonprotocol treatment will be left up to the treating physician if patient has an aMOI; waiting periods as described will apply
* ELIGIBILITY CRITERIA FOR THIRD SCREENING (STEP 4)
* Patient's disease has progressed on step 3 treatment or patient could not tolerate assigned treatment

  * Patient must meet one of the following criteria:

    * No response and progression (or inability to tolerate further treatment) occurred < 6 months from start of step 3 (second) treatment AND a biopsy was performed at step 2 screening

      * NOTE: Patients meeting these criteria will NOT be biopsied at this time point; instead, their latest MATCH assay results will be re-interrogated to determine if another treatment is available upon registration to this study step; it is not necessary to confirm the availability of another potential treatment assignment in advance OR
    * Progression (or inability to tolerate further treatment) occurred on step 3 treatment and a biopsy was not performed at step 2 screening (due to presence of a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6452 (Estimated)
Dates: Start 2015-08-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 90% two-sided confidence interval is calculated for ORR. For the purposes of this study, patients should be re-evaluated for response:
  * For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment on that step until death, or censored at the date of last contact, assessed up to 3 years
  Will be evaluated specifically for each drug (or step). OS will be estimated using the Kaplan-Meier method.
6-month progression free survival (PFS) rate | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed at 6 months
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Progression free survival | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed up to 3 years
  PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Keith T Flaherty, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1414):
- United States (1409):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - City of Hope Corona, Corona, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Pacific Cancer Care-Monterey, Monterey, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Saint Joseph's Medical Center, Stockton, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - City of Hope West Covina, West Covina, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - Broward Health North, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Health Central, Ocoee, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - The Longstreet Clinic - Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Newman Regional Health, Emporia, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Saint Elizabeth Healthcare Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - The NeuroMedical Center-Clinic, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Ochsner Medical Center West Bank, Gretna, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - New England Cancer Specialists - Kennebunk, Kennebunk, Maine
  - MaineHealth Stephens Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - New England Cancer Specialists - Topsham, Topsham, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - MetroWest Medical Center-Framingham Union Hospital, Framingham, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Hematology Oncology - Hayes, Clinton Township, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Michigan State University, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Carolina Surgical - Randolph, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Redeemer Health, Meadowbrook, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Suburban Community Hospital and Cancer Center, Norristown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Nazareth Hospital, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Oncology Hematology Association, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Newport Hospital, Newport, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Integrity Oncology PLLC-Collierville, Collierville, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - Covenant Health Cancer Centers, Knoxville, Tennessee
  - Covenant Health Cancer Centers - West, Knoxville, Tennessee
  - Covenant Health Oncology Group - Maryville, Maryville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Covenant Health Oncology Group - Oak Ridge, Oak Ridge, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Memorial Hermann Northeast Hospital, Humble, Texas
  - MD Anderson League City, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Memorial Hermann The Woodlands Hospital, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam
- Puerto Rico (4):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Tsao AS, Song Z, Ho AL, Mehnert JM, Ivy P, Gray RJ, Wang V, McShane LM, Rubinstein LV, Patton DR, Williams PM, Hamilton SR, Takebe N, Ajumally R, Silhavy J, Rahmanian S, Das B, Chen L, Karlovich C, Lococo JS, Tricoli JV, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of Vismodegib in Patients With SMO- or PTCH1-Mutated Tumors: Results From the National Cancer Institute Molecular Analysis for Therapy Choice Eastern Cooperative Oncology Group-American College of Radiology Imaging Network Trial (EAY131) Subprotocol T. JCO Precis Oncol. 2025 Oct;9:e2500119. doi: 10.1200/PO-25-00119. Epub 2025 Oct 9. PMID 41066729
- [Derived] Janku F, Jegede OA, Puhalla SL, Konstantinopoulos PA, Meric-Bernstam F, Zwiebel JA, Gray RJ, Wang XV, McShane LM, Rubinstein LV, Patton DR, Williams PM, Hamilton SR, Takebe N, Ghani S, Tricoli JV, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. PIK3CB Inhibitor GSK2636771 in Cancers With PTEN Mutation/Deletion or Loss of PTEN Protein Expression: Results From the NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocols N and P. JCO Precis Oncol. 2025 Aug;9:e2500265. doi: 10.1200/PO-25-00265. Epub 2025 Aug 27. PMID 40865033
- [Derived] Gouda MA, Wei Z, Rodon J, Davies MA, Janku F, Gray RJ, Wang V, McShane LM, Rubinstein LV, Patton DR, Williams PM, Hamilton SR, Liu R, Bota DA, Swiecicki PL, Buchschacher GL, Tricoli JV, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of Copanlisib in Patients With PTEN Loss: Results From NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocols Z1G and Z1H. JCO Precis Oncol. 2025 Feb;9:e2400451. doi: 10.1200/PO-24-00451. Epub 2025 Feb 6. PMID 39913886
- [Derived] Gien LT, Song Z, Poklepovic A, Collisson EA, Zwiebel JA, Gray RJ, Wang V, McShane LM, Rubinstein LV, Patton DR, Williams PM, Hamilton SR, Tricoli JV, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of Sunitinib in Tumors With c-KIT Mutations: Results From the NCI MATCH ECOG-ACRIN Trial (EAY131) Subprotocol V. JCO Precis Oncol. 2024 Dec;8:e2400514. doi: 10.1200/PO-24-00514. Epub 2024 Dec 12. PMID 39666929
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] O'Dwyer PJ, Gray RJ, Flaherty KT, Chen AP, Li S, Wang V, McShane LM, Patton DR, Tricoli JV, Williams PM, Iafrate AJ, Sklar J, Mitchell EP, Takebe N, Sims DJ, Coffey B, Fu T, Routbort M, Rubinstein LV, Little RF, Arteaga CL, Marinucci D, Hamilton SR, Conley BA, Harris LN, Doroshow JH. The NCI-MATCH trial: lessons for precision oncology. Nat Med. 2023 Jun;29(6):1349-1357. doi: 10.1038/s41591-023-02379-4. Epub 2023 Jun 15. PMID 37322121
- [Derived] Wisinski KB, Flamand Y, Wilson MA, Luke JJ, Tawbi HA, Hong F, Mitchell EP, Zwiebel JA, Chen H, Gray RJ, Li S, McShane LM, Rubinstein LV, Patton D, Williams PM, Hamilton SR, Behrens RJ, Pennington KP, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Trametinib in Patients With NF1-, GNAQ-, or GNA11-Mutant Tumors: Results From the NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocols S1 and S2. JCO Precis Oncol. 2023 Apr;7:e2200421. doi: 10.1200/PO.22.00421. PMID 37053535
- [Derived] Schrottmaier WC, Kral-Pointner JB, Salzmann M, Mussbacher M, Schmuckenschlager A, Pirabe A, Brunnthaler L, Kuttke M, Maier B, Heber S, Datler H, Ekici Y, Niederreiter B, Heber U, Blomgren B, Gorki AD, Soderberg-Naucler C, Payrastre B, Gratacap MP, Knapp S, Schabbauer G, Assinger A. Platelet p110beta mediates platelet-leukocyte interaction and curtails bacterial dissemination in pneumococcal pneumonia. Cell Rep. 2022 Nov 8;41(6):111614. doi: 10.1016/j.celrep.2022.111614. PMID 36351402
- [Derived] Krop IE, Jegede OA, Grilley-Olson JE, Lauring JD, Mitchell EP, Zwiebel JA, Gray RJ, Wang V, McShane LM, Rubinstein LV, Patton D, Williams PM, Hamilton SR, Kono SA, Ford JM, Garcia AA, Sui XD, Siegel RD, Slomovitz BM, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of Taselisib in PIK3CA-Mutated Solid Tumors Other Than Breast and Squamous Lung Cancer: Results From the NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocol I. JCO Precis Oncol. 2022 Feb;6:e2100424. doi: 10.1200/PO.21.00424. PMID 35138919
- [Derived] Damodaran S, Zhao F, Deming DA, Mitchell EP, Wright JJ, Gray RJ, Wang V, McShane LM, Rubinstein LV, Patton DR, Williams PM, Hamilton SR, Suga JM, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of Copanlisib in Patients With Tumors With PIK3CA Mutations: Results From the NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocol Z1F. J Clin Oncol. 2022 May 10;40(14):1552-1561. doi: 10.1200/JCO.21.01648. Epub 2022 Feb 8. PMID 35133871
- [Derived] Flaherty KT, Gray RJ, Chen AP, Li S, McShane LM, Patton D, Hamilton SR, Williams PM, Iafrate AJ, Sklar J, Mitchell EP, Harris LN, Takebe N, Sims DJ, Coffey B, Fu T, Routbort M, Zwiebel JA, Rubinstein LV, Little RF, Arteaga CL, Comis R, Abrams JS, O'Dwyer PJ, Conley BA; NCI-MATCH team. Molecular Landscape and Actionable Alterations in a Genomically Guided Cancer Clinical Trial: National Cancer Institute Molecular Analysis for Therapy Choice (NCI-MATCH). J Clin Oncol. 2020 Nov 20;38(33):3883-3894. doi: 10.1200/JCO.19.03010. Epub 2020 Oct 13. PMID 33048619
- [Derived] Chae YK, Hong F, Vaklavas C, Cheng HH, Hammerman P, Mitchell EP, Zwiebel JA, Ivy SP, Gray RJ, Li S, McShane LM, Rubinstein LV, Patton D, Williams PM, Hamilton SR, Mansfield A, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of AZD4547 in Patients With Tumors Harboring Aberrations in the FGFR Pathway: Results From the NCI-MATCH Trial (EAY131) Subprotocol W. J Clin Oncol. 2020 Jul 20;38(21):2407-2417. doi: 10.1200/JCO.19.02630. Epub 2020 May 28. PMID 32463741
- [Derived] Moore KN, Mannel RS. Is the NCI MATCH trial a match for gynecologic oncology? Gynecol Oncol. 2016 Jan;140(1):161-6. doi: 10.1016/j.ygyno.2015.11.003. Epub 2015 Nov 14. PMID 26586415
- See also: Related Info — https://www.cancer.gov/about-cancer/treatment/clinical-trials/nci-supported/nci-match

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT02465060/Prot_SAP_000.pdf